CLINICAL TRIAL: NCT05351411
Title: The Effect of Combined Progressive Functional Exercise on Contactin-1 and Contactin-2 Level in Mildly Disabled Persons With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Exercise on Contactin-1 and Contactin-2 Level in Persons With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, Lecturer, Firat University
Other Study IDs: FıratUniversit
Record Dates: First submitted 2022-04-16; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; exercise; contactin 1; contactin 2
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- combined progressive functional exercise: The initial implementation for the 8-week (3 days per week) combined exercise program consisted of a progressive aerobic exercise program with a lower extremity bike. The second part of the combined exercise program, the progressive resistance training program, is designed to be consistent with the resistance training section of the Canadian Physical Activity Guidelines for adults with MS. Each prescribed session consisted of 1-3 sets and 10-15 repetitions of 10 exercises targeting major muscle groups of the upper and lower extremities. The specific exercises prescribed included lunges, chair raises/squats, calf raises, knee flexion, knee extensions, shoulder rows, shoulder lateral raises, elbow flexions, elbow extensions, and abdominal curls.
- Placebo: Participants in the control group maintained their routine and had the opportunity to take part in the combined progressive functional exercise intervention after follow-up assessments had been conducted.

INTERVENTIONS:
Other:  — Participants in the control group maintained their therapeutic routine and had the opportunity to take part in the combined progressive functional exercise intervention after follow-up assessments had been conducted.
  Groups: combined progressive functional exercise

SUMMARY:
Little is known about the potential effects of exercise on the underlying disease mechanisms in multiple sclerosis (MS). Although contactin-1 and contactin-2 are known as two proteins involved in axonal regeneration, it is unclear whether these proteins are induced by exercise in persons with MS (PwMS). The aim of this study was to determine the serum levels of contactin-1 and contactin-2 in PwMS and to investigate the change of these markers with exercise. Although contactin-1 and contactin-2 are known as two proteins involved in axonal regeneration, the mechanism of action of these proteins in MS patients has not been fully elucidated in the literature. The investigators' aim was to determine the serum levels of contactin-1 and contactin-2 in a group of relapsing-remitting multiple sclerosis (RRMS) patients and to evaluate the change of these markers with exercise. Thus, the investigators think that a valuable contribution will be made to the literature to shed light on the role of biomarkers in the mechanism mediating the beneficial effects of exercise in MS. In addition, as far as the investigators know, this study is the first to investigate the effect of exercise on contactin-1 and contactin-2 serum levels in MS patients.

DETAILED DESCRIPTION:
This randomized controlled trial with a blinded outcome assessment evaluated an 8-week (3 sessions per week) training intervention to determine the effect of exercise on contactin-1 and contactin-2 in persons with RRMS. The participants were divided into the intervention and control groups by stratified randomization. Stratification was randomly assigned as 1≤ EDSS ≤ 3 and 3< EDSS ≤5.5 using Windows-based SPSS 25.0. (SPSS Inc., Chicago, Illinois, USA). All measurements and tests were performed before and after the 8-week exercise program. Blood samples were taken for analysis of contactin-1 and contactin-2 serum levels, after which participants completed a cognitive performance and a cardiopulmonary exercise test.

The current study was approved by the Fırat University Human Research Ethics Local Committee (2021/12-38) and was conducted in accordance with the Declaration of Helsinki. All participants were informed about the study and their written informed consent was obtained before the study. Participants performed a graded cardiopulmonary exercise test on a cycle ergometer (Ergoline Ergoselect 200; Ergoline GMBH, Bitz, Germany) at the beginning to determine their maximum aerobic capacity. The test was stopped at the moment of voluntary exhaustion, when patients were unable to maintain cadence (<50 rpm), the maximum effort was achieved, or for safety reasons. Venous blood was drawn using venipuncture and clotted for serum and centrifuged at 4000g for 5 minutes at 4°C. Serum samples then were aliquoted, and stored at -80°C until were assayed with enzyme-linked immunosorbent assay (ELISA) analysis. The serum levels of Contactin-1 (Cat.No: E-EL-H1498) and Contactin-2 (Cat.No: E-EL-H1499) were measured with commercially available specific human ELISA kits (Elabscience, Houston, Texas, United States). Paced Auditory Serial Addition Test with the 3-second stimulus (PASAT-3) was used as a measure of cognitive performance including information processing speed, working memory and sustained attention

ELIGIBILITY:
Inclusion Criteria:

* definite diagnosis of RRMS according to the McDonalds criteria,
* 18 years or older,
* EDSS levels of 1.0 - 5.5, EDSS "pyramidal functions" sub score ≥2,
* who have not had an attack in the last 3 months,
* who were patients who did not receive steroid treatment for the last 3 months.

Exclusion Criteria:

* orthopedic, cardiopulmonary, or systemic problems that prevent participation in exercises,
* pregnancy,
* started immunomodulatory treatment in the last 6 months,
* participated in resistance training 3 months before inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out on individuals with MS followed in the Neurology Clinic of Fırat University Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Biomarker - Contactin 1 | 8 weeks
  Venous blood was drawn using venipuncture and clotted for serum and centrifuged at 4000g for 5 minutes at 4°C. Serum samples then were aliquoted, and stored at -80°C until were assayed with enzyme-linked immunosorbent assay (ELISA) analysis.
Biomarker - Contactin 2 | 8 weeks
  Venous blood was drawn using venipuncture and clotted for serum and centrifuged at 4000g for 5 minutes at 4°C. Serum samples then were aliquoted, and stored at -80°C until were assayed with enzyme-linked immunosorbent assay (ELISA) analysis.

SECONDARY OUTCOMES:
Paced Auditory Serial Addition Test with 3-second stimulus (PASAT-3) | 8 weeks
  Paced Auditory Serial Addition Test with 3-second stimulus (PASAT-3) was used as a measure of cognitive performance including information processing speed, working memory and sustained attention

CONTACTS AND LOCATIONS:
Overall Officials: Caner F Demir, MD professor, Study Director — Firat University
Locations (1):
- Fırat university, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson AJ, Baranzini SE, Geurts J, Hemmer B, Ciccarelli O. Multiple sclerosis. Lancet. 2018 Apr 21;391(10130):1622-1636. doi: 10.1016/S0140-6736(18)30481-1. Epub 2018 Mar 23. PMID 29576504
- [Background] Negaresh R, Motl RW, Zimmer P, Mokhtarzade M, Baker JS. Effects of exercise training on multiple sclerosis biomarkers of central nervous system and disease status: a systematic review of intervention studies. Eur J Neurol. 2019 May;26(5):711-721. doi: 10.1111/ene.13929. Epub 2019 Mar 14. PMID 30734989
- [Background] Sandroff BM, Richardson EV, Motl RW. The Neurologist as an Agent of Exercise Rehabilitation in Multiple Sclerosis. Exerc Sport Sci Rev. 2021 Oct 1;49(4):260-266. doi: 10.1249/JES.0000000000000262. PMID 34049322
- [Background] Motl RW, Sandroff BM. Exercise as a Countermeasure to Declining Central Nervous System Function in Multiple Sclerosis. Clin Ther. 2018 Jan;40(1):16-25. doi: 10.1016/j.clinthera.2017.12.001. Epub 2017 Dec 26. PMID 29287750
- [Background] Schutzer SE, Angel TE, Liu T, Schepmoes AA, Xie F, Bergquist J, Vecsei L, Zadori D, Camp DG 2nd, Holland BK, Smith RD, Coyle PK. Gray matter is targeted in first-attack multiple sclerosis. PLoS One. 2013 Sep 10;8(9):e66117. doi: 10.1371/journal.pone.0066117. eCollection 2013. PMID 24039694
- [Result] Derfuss T, Parikh K, Velhin S, Braun M, Mathey E, Krumbholz M, Kumpfel T, Moldenhauer A, Rader C, Sonderegger P, Pollmann W, Tiefenthaller C, Bauer J, Lassmann H, Wekerle H, Karagogeos D, Hohlfeld R, Linington C, Meinl E. Contactin-2/TAG-1-directed autoimmunity is identified in multiple sclerosis patients and mediates gray matter pathology in animals. Proc Natl Acad Sci U S A. 2009 May 19;106(20):8302-7. doi: 10.1073/pnas.0901496106. Epub 2009 Apr 28. PMID 19416878
- [Result] Shimoda Y, Watanabe K. Contactins: emerging key roles in the development and function of the nervous system. Cell Adh Migr. 2009 Jan-Mar;3(1):64-70. doi: 10.4161/cam.3.1.7764. Epub 2009 Jan 6. PMID 19262165
- [Result] Colakoglu G, Bergstrom-Tyrberg U, Berglund EO, Ranscht B. Contactin-1 regulates myelination and nodal/paranodal domain organization in the central nervous system. Proc Natl Acad Sci U S A. 2014 Jan 21;111(3):E394-403. doi: 10.1073/pnas.1313769110. Epub 2014 Jan 2. PMID 24385581
- [Result] Dalgas U, Ingemann-Hansen T, Stenager E. Physical Exercise and MS Recommendations. Int MS J. 2009 Apr;16(1):5-11. PMID 19413920
- [Result] Ocklenburg S, Gerding WM, Arning L, Genc E, Epplen JT, Gunturkun O, Beste C. Myelin Genes and the Corpus Callosum: Proteolipid Protein 1 (PLP1) and Contactin 1 (CNTN1) Gene Variation Modulates Interhemispheric Integration. Mol Neurobiol. 2017 Dec;54(10):7908-7916. doi: 10.1007/s12035-016-0285-5. Epub 2016 Nov 18. PMID 27864734